CLINICAL TRIAL: NCT04540757
Title: ImPact on QualIty Of Life From Multi-modality Treatment for Lung caNcEr: A Randomised Controlled fEasibility tRial of Surgery Versus no Surgery as Part of Multi-modality Treatment in Potentially Resectable Stage III-N2 NSCLC (The PIONEER Trial)
Brief Title: Impact on Quality of Life From Multi-modality Lung Cancer
Acronym: PIONEER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp176
Record Dates: First submitted 2020-04-06; First posted 2020-09-07 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Lung Neoplasms; Quality of Life
Keywords: non small cell lung cancer; Stage III N2; Quality of life; Multi-modality treatment
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Surgery and systemic anti-cancer therapy (with or without radiotherapy) given in any order
  Interventions: Procedure: Surgery
- No surgery: Radiotherapy and systemic anti-cancer treatment given in any order (with or without adjuvant immunotherapy if indicated).
  Interventions: Procedure: No surgery

INTERVENTIONS:
Procedure: Surgery — Participants will be randomised to receive surgery as part of multi-modality treatment
  Groups: Surgery
Procedure: No surgery — Participants will be randomised to receive no surgery as part of multi-modality treatment
  Groups: No surgery

SUMMARY:
The investigators aim to explore how lung cancer patients and their family carers are affected by different types of cancer treatment. The investigators are focusing on a particular type of lung cancer called Stage III N2. N2 means the cancer has spread just outside the lung to the lymph nodes. There are two main treatments available in the UK for this type of lung cancer:

1. surgery PLUS chemo radiotherapy or chemotherapy
2. radiotherapy PLUS chemotherapy Patients live for a similar length of time with either treatment option so it is difficult for patients and health professionals to know which treatment to choose. It is important to understand the impact of the treatment on patients in their daily lives. Patients will be allocated at random to receive one of the two treatments options. Patients and carers will complete questionnaires and take part in interviews. The results of this study will help the investigators decide if a larger study should be conducted in the future.

DETAILED DESCRIPTION:
The investigators aim to explore how lung cancer patients and their family carers are affected by different types of cancer treatment.The information collected will help patients and their carers in the future to make decisions about the best treatment option for them. The investigators are focusing on a particular type of lung cancer called Stage III N2. N2 means the cancer has spread just outside the lung to the lymph nodes. Around 2500 patients a year in the UK are diagnosed with this type of lung cancer. There are two main treatments available in the UK:

1. surgery PLUS chemo radiotherapy or chemotherapy
2. radiotherapy PLUS chemotherapy Patients live for a similar length of time with either treatment option so it is difficult for patients and health professionals to know which treatment to choose. Research has not explored how the two different treatments offered affect individual patients and their carer. It is important to understand the impact of the treatment on:

   * Symptoms
   * Side effects
   * Emotional well-being
   * Day to day activities

Other research studies including N2 lung cancer patients have struggled with patient recruitment. This study design will show us if it is possible to run this type of research with this group of patients. Patients will be allocated at random to receive one of the two treatments options: 1) surgery PLUS chemo radiotherapy or chemotherapy 2) radiotherapy PLUS chemotherapy Patients and carers will complete questionnaires and take part in interviews. Health professionals will also be asked to take part in interviews. These interviews will help the investigators to understand their experience of recruiting patients to this study. The results of this study will help the investigators decide if a larger study should be conducted in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with potentially resectable T1-4 N2 M0 NSCLC who have received an multi disciplinary team recommendation for multi-modality treatment
* Multi disciplinary team consensus that the patient has adequate physiological reserve for multi-modality treatment and either treatment arm is both technically and clinically appropriate
* Patient over the age of 18 years

Carer criteria:

* Carers of patients who have consented to take part in the randomised controlled trial
* Over the age of 18 years

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients who are not able to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III N2 non small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Patients with N2 disease | 20 months
  Determine the proportion of patients with potentially resectable stage III N2 disease who are fit for surgery
Recruitment | 20 months
  Number of eligible patients recruited
Attrition | 26 months
  Number of patients lost to follow up
Treatment completion | 6 months
  The proportion of patients who complete their allocated treatment
Quality of life | 6 months
  Collected using the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30)
Quality of life | 6 months
  Collected using the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30-LC13)
Quality of life | 6 months
  Short Form 36 (SF36)
Anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale (HADS)
EuroQOL 5D | 6 months
  Quality of life (EQ5D)
Service use/health economics | 6 months
  Study specific service use and health economics questionnaire
Mortality rates | 6 months
  Mortality rates collected by clinicians

SECONDARY OUTCOMES:
Patient experience | 26 months
  Interviews will be conducted with patients to explore their experiences in more detail.
Carer quality of life | 6 months
  Carer Quality of life- cancer questionnaire
Caregiver burden | 6 months
  Zarit Caregiver Burden
Caregiver anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Manchester University Foundation Trust- Wythenshawe, Manchester

REFERENCES:
- [Derived] Taylor S, Yorke J, Tsim S, Navani N, Baldwin D, Woolhouse I, Edwards J, Grundy S, Robson J, Rhodes S, Gomes F, Blackhall F, Faivre-Finn C, Evison M. Impact on quality of life from multimodality treatment for lung cancer: a randomised controlled feasibility trial of surgery versus no surgery as part of multimodality treatment in potentially resectable stage III-N2 NSCLC (the PIONEER trial). BMJ Open Respir Res. 2021 Jul;8(1):e000846. doi: 10.1136/bmjresp-2020-000846. PMID 34266853